CLINICAL TRIAL: NCT06092294
Title: Effects of a Numerical Superiority and Numerical Inferiority Tactical Training Program Compared With Conventional Training on Procedural Tactical Knowledge and Executive Functions in Soccer Players
Brief Title: Numerical Superiority and Inferiority Compared With Conventional Training on PTK and Executive Functions in Soccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Club La Nororiental (Unknown)
Responsible Party: Principal Investigator, Juan Osvaldo Jiménez Trujillo, Magister, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Procedural Tactical Knowledge
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Decision Making in Soccer Players and Executive Functions
Keywords: Competence in Soccer Players; Decision Making; Executive Functions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study has masking at 2 levels. the first one is in the outcome assessors and the second level of masking is in the analysis of the data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tactical training in numerical superiority and numerical inferiority (Experimental): Participants will carry out a specific training program, with the objective of improving both offensive and defensive Tactical-Technical Actions (ATT) that will allow the increase of effectiveness indexes (EI) (offensive and defensive). The formats through which will train are Small Sided Games (SSGs) and ATT 2 against 1, 3 against 2 and 4 against 3 alternating them during the week (SSGs on Tuesdays and ATT on Thursdays).
  The characteristics of this training program are: training frequency 5 times/week, plus 1 competition on weekends, frequency of stimulation of the SSGs and ATT of numerical superiority and numerical inferiority 2 times/week, the specific training time assigned to the development of these formats and exercises will be 30 to 42 minutes/training session and will be carried out after the warm-up.
  Interventions: Behavioral: Tactical training in numerical superiority and numerical inferiority
- Conventional training in numerical equality (Active Comparator): On the other hand, the CG participants will perform conventional training. In the present study, conventional training is defined as ATTs performed in equal numbers in 1 against 1, 2 against 2 and 3 against 3 formats. Likewise, coaches will be asked not to carry out additional specific training with these formats, nor of SSGs or offensive or defensive ATT in numerical superiority and inferiority, specifically in 2 against 1, 3 against 2, or 4 against 3 formats, during the time of the study, to avoid confusion biases due to possible co-interventions. This CG training program will include individual, couples, and groups of three ATTs .
  The characteristics of this training program are: training frequency 5 times/week, 1 official competition on weekends, frequency of ATT stimulation in 1v1, 2v2 and 3v3 formats is 2 times/week, the specific training time allocated will be 40 minutes per training session and will be performed after the warm-up.
  Interventions: Behavioral: Conventional training in numerical equality

INTERVENTIONS:
Behavioral: Tactical training in numerical superiority and numerical inferiority — In the present study, the SSGs training sessions will be carried out in the following areas:
  2c1: length 11.5m and width 9m (total: 103.5m2), equivalent to 34.5m2 for each player.
  3c2: length 14m and width 12m (total: 168m2), equivalent to 33.6m2 for each player.
  4c3: length 17m and width 14m (total: 238m2), equivalent to 34m2 per each player.
  Arms: Tactical training in numerical superiority and numerical inferiority
Behavioral: Conventional training in numerical equality — Coach who will run the CG training program will be different from the coach who will run the GE training program. As with the GE, a coach will also be assigned to the CG to record, quantify and monitor the training stimuli of this comparison group, who will record it on forms designed for this purpose.
  Arms: Conventional training in numerical equality

SUMMARY:
There is a great need to establish reliable evaluation and intervention protocols to improve the tactical component, decision making (DM) and procedural tactical knowledge (PTK) in soccer. Objectives: to determine the effects of a 12-week follow up numerical superiority and numerical inferiority tactical training program on PTK, which will be evaluated by calculating offensive, defensive and global effectiveness indexes (EI) of 24 amateur male soccer players, as well as the effect on their executive functions. Method: randomized controlled trial, with two groups in parallel, experimental group (EG) and control group (CG), with different measurements over time (pretest, intermediate test 1, intermediate test 2 and posttest).

DETAILED DESCRIPTION:
Program characteristics: training frequency 5 times/week, 1 competition, frequency of stimulation of small side games (SSGs) and technical-tactical actions (ATT) of numerical superiority and inferiority 2 times/week, specific training time 30 to 42 minutes/session. The PTK will be evaluated through the Football Competence Observation System (FOCOS). Data analysis: Shapiro-Wilk will be applied and according to the results, the data will be summarized with means and standard deviation or with medians and interquartile ranges. A repeated measures design will be performed using ANOVA and MANOVA will also be performed. In addition, the assumption of homogeneity of the variances will be evaluated based on the Levene statistics. For executive functions, intragroup analysis will be performed using dependent Student's t-test or Wilcoxon. For intergroup analysis, t student for independent samples or U Mann Withney will be applied. Confidence intervals (CI95) and effect sizes for two tails will be reported, with an alpha (α) set at 0.05 and statistical power of 0.8 (1-β). Statistical significance (p≤0.05). SPSS version 27 and R version 4.0 will be used. Ethical aspects: the guidelines of the Declaration of Helsinki (2013) and the Ministry of Health and Social Protection (resolution 8430/1993) will be followed, this research is of minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players belonging to a soccer club.
* Who play the role of field players (all except goalkeepers).
* Who compete in the First B category of the Antioquia Soccer League in the 2023 season.
* Players between 17 and 26 years of age.
* Players with at least six months of experience in federated soccer.
* Players who do not present cognitive disorders that hinder learning, which can be identified through monitoring by coaches and/or tests conducted by the Neuropsychology staff.
* They must be affiliated to the contributory or subsidized health system.
* They must agree to participate in the study after knowing and signing the informed consent or assent, as appropriate.

Exclusion Criteria:

* Players with musculoskeletal disorders at the time of sample selection.
* Players recovering from injury.

Ages: 17 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Offensive Effectiveness Index (OEI). Scale for measuring the OEI ranges from 0 to 1 (0 being the worst score and 1 being the best score). These scores will be obtained by video analysis of 21 soccer players' tactical behaviors by the video analyst | 16 weeks
  The OEI is determined through the following formula:
  OEI = Volume of successful tactical behaviors/Number of tactical behaviors developed in each category of analysis.
  OEI = Sum of the EI of the offensive tactical behaviors/Number of categories in which the player developed offensive tactical behaviors.

SECONDARY OUTCOMES:
Defensive Effectiveness Index (DEI). Scale for measuring the DEI ranges from 0 to 1 (0 being the worst score and 1 being the best score). These scores will be obtained by video analysis of 10 soccer players' tactical behaviors by the video analyst. | 16 weeks
  The DEI is determined through the following formula:
  DEI = Volume of successful tactical behaviors/Number of tactical behaviors developed in each category of analysis.
  DEI = Sum of the EI of the defensive tactical behaviors/Number of categories in which the player developed defensive tactical behaviors.

OTHER OUTCOMES:
Executive Functions Measurements will be evaluated according to the number of hits and errors and the time taken to complete the evaluations (the better the one who presents more hits, fewer errors and performs the tests in the shortest time) | 16 weeks
  Executive functions is a term used to describe cognitive processes that regulate thought and action such as problem solving, planning, sequencing, sustained and selective attention, inhibition, use of feedback, multitasking, cognitive flexibility and ability to deal with novel situations.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Osvaldo Jimenez Trujillo, Principal Investigator — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT06092294/Prot_SAP_000.pdf